CLINICAL TRIAL: NCT07004673
Title: 18F FDG and 68Ga FAPI PET/MR Imaging of Carotid Artery Plaque Vulnerability: A Clinical Study in Carotid Artery Plaque Patients
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: 18F FDG and 68Ga FAPI PET/MR
Record Dates: First submitted 2025-04-21; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-04

CONDITIONS: Carotid Artery Plaque; Ischemic Stroke; PET / MR
MeSH Terms: conditions — Carotid Stenosis; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carotid plaque & carotid atherosclerotic stenosis: Medication or carotid stenting or carotid endarterectomy according to clinical guidelines

SUMMARY:
Carotid atherosclerotic plaque rupture is the main cause of ischemic stroke attacks, and early and precise assessment of plaque vulnerability can prevent ischemic stroke. High-resolution MRI can reflect vulnerable plaque features such as thin fibrous caps and large lipid cores, but cannot assess their metabolic information; Fibro-activated proteins (FAPs) of PET are specifically expressed in atherosclerosis and suggest vulnerable plaques by reflecting inflammation-induced fibrosis. The aim of this study was to apply 18F FDG&68Ga-FAPI PET/MR imaging to investigate the vulnerability of carotid atherosclerotic plaques, to obtain quantitative evaluation indexes of active fibrosis within carotid plaques, and to clarify the PET/MR characteristics of unstable plaques in carotid arteries

ELIGIBILITY:
Inclusion Criteria:

-Age between 18 and 80 years; Presence of carotid atherosclerotic plaque confirmed by ultrasound within the past two weeks, with carotid intima-media thickness (IMT) ≥ 2 mm (IMT ≥ 1.2 mm is defined as carotid atherosclerosis) or carotid artery stenosis ≥ 50% as indicated by CTA.

Exclusion Criteria:

* Absolute or relative contraindications related to PET/MR imaging safety (e.g., metallic implants, MRI phobia, etc.); Patients who have undergone carotid endarterectomy (CEA) or carotid artery stenting (CAS); Pregnant or lactating women; Presence of other vascular diseases, such as vasculitis, moyamoya disease, arterial dissection, etc.; Severe agitation or inability to cooperate with imaging procedures.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study included a total of 100 patients with internal carotid artery atherosclerosis, divided into 50 cases in the symptomatic group and 50 cases in the asymptomatic group.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
stroke from baseline to 1months after PET/MR | 1 month after PET/MRI
  1. Incidence of ipsilateral carotid cerebral infarction Incidence within 1 month of standard drug therapy or carotid stenting or carotid endarterectomy
stroke from baseline to 6 months after PET/MR | 6 month after PET/MRI
  1. Incidence of ipsilateral carotid cerebral infarction Incidence within 6 month of standard drug therapy or carotid stenting or carotid endarterectomy
stroke from baseline to 12 months after PET/MR | 12 month after PET/MRI
  1. Incidence of ipsilateral carotid cerebral infarction Incidence within 12 month of standard drug therapy or carotid stenting or carotid endarterectomy
cerebral hemorrhage from baseline to 1months after PET/MR | 1 month after PET/MRI
  1. Incidence of ipsilateral carotid cerebral hemorrhage Incidence within 1 month of standard drug therapy or carotid stenting or carotid endarterectomy
Lumen patency rate of ipsilateral carotid artery from baseline to 1 months after PET/MR | 1 month after PET/MRI
  1、The rate of ipsilateral carotid artery lumen patency Observe the rate of lumen patency within 1 month after standard drug therapy or carotid stenting or carotid endarterectomy.
Lumen patency rate of ipsilateral carotid artery from baseline to 6 months after PET/MR | 6 month after PET/MRI
  1、The rate of ipsilateral carotid artery lumen patency Observe the rate of lumen patency within 6 month after standard drug therapy or carotid stenting or carotid endarterectomy.
Lumen patency rate of ipsilateral carotid artery from baseline to 12 months after PET/MR | 12 month after PET/MRI
  1、The rate of ipsilateral carotid artery lumen patency Observe the rate of lumen patency within 12 month after standard drug therapy or carotid stenting or carotid endarterectomy.

SECONDARY OUTCOMES:
18F FDG and 68Ga FAPI PET-MRI imaging results from baseline to 1 months after PET/MRI | 1month after PET/MRI
  1. Changes in metabolic rate of ipsilateral carotid plaque Changes in metabolic rate of 18F FDG and 68Ga FAPI within 1 month after standard drug therapy or carotid stenting or carotid endarterectomy were observed
18F FDG and 68Ga FAPI PET-MRI imaging results from baseline to 6 months after PET/MRI | 6 month after PET/MRI
  1. Changes in metabolic rate of ipsilateral carotid plaque Changes in metabolic rate of 18F FDG and 68Ga FAPI within 6 month after standard drug therapy or carotid stenting or carotid endarterectomy were observed
18F FDG and 68Ga FAPI PET-MRI imaging results from baseline to 12 months after PET/MRI | 12 month after PET/MRI
  1. Changes in metabolic rate of ipsilateral carotid plaque Changes in metabolic rate of 18F FDG and 68Ga FAPI within 12 month after standard drug therapy or carotid stenting or carotid endarterectomy were observed

CONTACTS AND LOCATIONS:
Overall Officials: Jun Liu Jun Liu, Study Chair — Department of Neurology, Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine Study Chair
Locations (1):
- Department of neurology, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No